CLINICAL TRIAL: NCT02415725
Title: Early Detection of Secondary Lymphedema After Cancer Treatments
Brief Title: Early Detection of Lymphedema After Cancer Treatments
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire Saint Pierre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2LEED-ICG
Record Dates: First submitted 2015-03-27; First posted 2015-04-14 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-03

CONDITIONS: Lymphadenectomy; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- lymphofluoroscopy (Experimental): Indocyanine Green intradermal injection before surgery, and after 3, 6 and 12 monthes
  Interventions: Drug: Indocyanine Green

INTERVENTIONS:
Drug: Indocyanine Green — visualization of the architecture of superficial lymphatic network after Indocyanine Green injection
  Other Names: ICG

SUMMARY:
Many clinical situations in oncologic surgery imply the need to dissect more or less extensively lymph node stations which are in direct relation with the lymphatic drainage of the anatomical region affected by cancer.

The dissected lymph nodes drain generally several regions, and their dissection reduces then the drainage capacity of all these regions, increasing the risk for the patient to develop a secondary lymphedema, shorter or longer after surgery.

Efficient treatments exist, but are difficult to implement and to continue for a long time.The later the treatment of the lymphedema begins, the heavier it is, both on the medical and socio-economic level.

The lymphofluoroscopy, shows that some oncologic patients, operated and free of apparent secondary lymphedema, present abnormalities of the lymphatic network.

The present study aims to confirm that it is now possible to detect secondary lymphedema at a subclinical stage.

DETAILED DESCRIPTION:
Many clinical situations in oncologic surgery imply the need to dissect more or less extensively lymph node stations which are in direct relation with the lymphatic drainage of the anatomical region affected by cancer.

The dissected lymph nodes drain generally several regions, and their dissection reduces then the drainage capacity of all these regions, increasing the risk for the patient to develop a secondary lymphedema, shorter or longer after surgery.

The recent meta-analysis show that nearly 15% of patient operated for a cancer with lymph node dissection develop after 27 months from surgery a lymphedema of the limb corresponding to the operated region.

Radio- and chemotherapy may especially encumber the already reduced lymphatic capacity.

The impact on the health and the quality of life of the patient is very significant on the physical and psychological aspect, but also on social and economic aspect.

Efficient treatments exist, but are difficult to implement and to continue for a long time. They are considered as serious diseases which are expensive for the INAMI. Lymphedema is a chronic disease which needs repeated and continued treatments. The later the treatment of the lymphedema begins, the heavier it is, both on the medical and socio-economic level. Some patients even lose their job because of their functional infirmity.

Here the investigators remind that lymphedema is painless, even in its most spectacular cases.

Still currently, a lymphedema is diagnosed after it has developed, and only when the functional discomfort, or the physical appearance disturb the patient enough to go to consultation.

The lymphofluoroscopy (new emerging imaging technique in the field of lymphology) used since 3 years by the promoters of the present project, shows that some oncologic patients, operated and free of apparent secondary lymphedema, present abnormalities of the lymphatic network. These patients report heaviness sensations or sporadic paraesthesia which generally does not arouse suspicion of beginning lymphedema.

The present prospective, multidisciplinary and multicentric clinical study aims to confirm that it is now possible to detect secondary lymphedema at a subclinical stage. In a second step, prevention will be considered. Detection may be performed using a simple lymphofluoroscopic examination, which is a minimally invasive and inexpensive imaging technique. It allows to realize a mapping of the superficial lymphatic network and to identify the characteristics of the secondary lymphedema in the group of patients at risk to develop lymphedema after lymph node dissection.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will undergo lymphadenectomy (either large lymphadenectomy or sentinel lymph node biopsy) for oncologic reason (gynaecologic, urologic or mammary cancer, melanoma and other skin cancer) without measurable or observable limb lymphedema.
* Informed consent form signed.

Exclusion Criteria:

* Allergy to iodine.
* Incapaciy to give informed consent.
* < 18 years.
* Pregnancy or breastfeeding.
* Coronary disease.
* Advanced renal impairment.
* Hyperthyroidism.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2014-09; Primary Completion 2017-12 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
number of lymphatic vessels visualized | 12 monthes

CONTACTS AND LOCATIONS:
Overall Officials: Liesbeth Vandermeeren, MD, Principal Investigator — CHU St-Pierre
Locations (1):
- CHU St-Pierre - Clinique de Lymphologie, Brussels, Belgium